CLINICAL TRIAL: NCT03165214
Title: Effectiveness of Embolization of Pelvic Veins in Treatment of Pelvic Congestion Syndrome
Brief Title: Embolization of Pelvic Veins in Treatment of Pelvic Congestion Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients recruited
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PCS
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Congestive Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coil group (Active Comparator): micro coils
  Interventions: Device: coil
- glue group (Experimental): hystoacryl mixed with lipidol
  Interventions: Device: hystoacryl glue

INTERVENTIONS:
Device: coil — microcoils
  Arms: coil group
Device: hystoacryl glue — hystoacryl mixed with lipidol
  Arms: glue group

SUMMARY:
Chronic pelvic pain is defined as chronic or persistent pain perceived in structures related to the pelvis of either men or women for more than 6 months according to The International Association for the Study of Pain. In other words, chronic pelvic pain with associated ovarian vein varicosities is termed pelvic congestion syndrome and is an important but under-diagnosed condition

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms of pelvic congestion syndrome documented by Doppler ultrasound
* Failed medical treatment.

Exclusion Criteria:

* Endometriosis.
* Uterine fibroids.
* Previous pelvic operations.
* Urological diseases.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
The number of treated patients with different interventions | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Assiut Faculty of Medicine, Asyut

IPD SHARING:
Plan to Share IPD: No